CLINICAL TRIAL: NCT01413997
Title: Feasibility Study of Connective Tissue Motion Measure - a Biomarker for Perimuscular Connective Tissue Pathology.
Brief Title: Connective Tissue Motion Measure
Acronym: CTMM1
Status: Completed | Type: Observational
Sponsor: Stromatec, Inc. (Industry)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Robert Davis, CEO, Stromatec, Inc.
Other Study IDs: ctmmp1-R43AT006085; 1R43AT006085-01 (NIH)
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chronic Low Back Pain
- No Low Back Pain

SUMMARY:
The goal of this project is to develop a biomarker - the Connective Tissue Motion Measure (CTMM) -quantifying the functional behavior of perimuscular connective tissues.

DETAILED DESCRIPTION:
The differential motion between specific connective tissue strata will be measured during tissue displacement (linear oscillation) initiated by a computer-controlled needle stimulus tool (NST). The CTMM will be suitable as an outcome measure for mechanistic and clinical studies of CAM interventions. The CTMM also will potentially serve as a clinical diagnostic and treatment-monitoring tool for manual therapists, acupuncturists, and CAM clinicians interested in assessing the functional status of a patient's connective tissue.

ELIGIBILITY:
Inclusion criteria for LBP subjects:

* history of recurrent or chronic LBP for a minimum of 12 months
* ability to stand and walk without assistance
* ability to understand and read English
* ability to understand and sign a consent form

Inclusion criteria for No-LBP subjects:

* no history of low back pain or any other chronic pain that has limited activities of daily living or work
* a numerical current pain index of less than 0.5.

Exclusion Criteria for all subjects:

* previous severe back or low extremity injury or surgery
* major structural spinal deformity (scoliosis, kyphosis, stenosis)
* ankylosing spondylitis or rheumatoid arthritis
* neurological deficit (weakness and/or sensory loss, decreased deep tendon reflexes suggesting nerve root compression, but not subjective symptoms of nerve root irritation (sciatica)
* neurological or major psychiatric disorder
* bleeding disorders
* corticosteroid or anticoagulant medication
* pregnancy
* worker's compensation or disability case
* in litigation for the LBP problem
* acute systemic infection
* BMI less than 21 or greater than 35

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stromatec, Inc., Burlington, Vermont, United States